CLINICAL TRIAL: NCT01289535
Title: Immune Response Analysis to Influenza Vaccine in Elderly Aged Over 65 Years
Acronym: Expand IDWP21
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010.621
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Immune Response
Keywords: Influenza vaccine; immune response; elderly
MeSH Terms: conditions — Influenza, Human | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- antibody rates (Experimental)
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Blood sample of 7 ml

SUMMARY:
This study is the first step in a clinical research program that aims to study the immune response to influenza vaccine in the elderly and then to propose a new method of administering the vaccine.

Influenza can cause severe complications in patients at risk (elderly and subjects vulnerable because of a chronic underlying disease). Over 90% of deaths related to influenza occur in people aged over 65 years.

Vaccination is the most effective way to prevent infection. The World Health Organization recommends annual immunization for people at risk, including all persons aged over 65 years, to reduce the risk of morbidity and mortality related to influenza.

However, the immune response to influenza vaccine appears to be lower in elderly than in young people.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 65 years or over
* Influenza vaccination without adjuvant, within 3 weeks and 3 months before inclusion visit
* Legal capacity to consent
* Subject had given written consent before his participation

Exclusion Criteria:

* Adjuvanted influenza vaccine (e.g: Fluad, Gripguard)
* Live vaccines within 3 weeks before and after influenza vaccination
* Inactivated vaccines within 2 weeks before and after influenza vaccination
* Chronic disease non-stabilized under treatment
* Severe malnutrition in the opinion of the investigator
* Congenital immunodeficiency
* Chemotherapy or radiotherapy over the last 6 months
* Immunosuppressive therapy or corticosteroid (daily dose of prednisone or equivalent >/= 20 mg/d over 14 days) from 1 month before vaccination until the study visit
* Participation in another clinical study that could interfere with the present study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
antibody rates after influenza vaccination | up to 3 months after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Recherche Clinique en Immunologie Lyon Sud (URCI-LS) et Service d'Immunologie clinique et allergologie, Pierre-Bénite, France